CLINICAL TRIAL: NCT00165347
Title: Phase II Study of PTK787/ZK222584 in Multiple Myeloma
Brief Title: Protein Tyrosine Kinases (PTK) in Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Brigham and Women's Hospital (Other); Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 03-257
Record Dates: First submitted 2005-09-09; First posted 2005-09-14 (Estimated); Last update posted 2007-12-21 (Estimated); Status verified 2007-12

CONDITIONS: Multiple Myeloma
Keywords: Multiple myeloma; PTK; Relapsed multiple myeloma; Refractory Multiple myeloma; Myeloma
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell | interventions — vatalanib

INTERVENTIONS:
Drug: PTK787/ZK222584

SUMMARY:
The purpose of this study is to determine whether or not cancer cells in the body are affected by PTK and whether it affects the growth of these cells.

DETAILED DESCRIPTION:
Patients will take PTK orally once a day for the duration of their time on the study. Each cycle of chemotherapy will last for 4 weeks.

Measurement of vital signs will be done weekly during the first month of treatment.

Physical exam, vital signs, blood work, a quality of life assessment, and x-ray or MRI wil be performed every 4 weeks.

Patients will remain on the study until their disease fails to respond to treatment or there are intolerable side effects. Typically treatment is performed for 12 weeks and up to one year in patients that are stable and responding.

ELIGIBILITY:
Inclusion Criteria:

* Older than 18 years of age.
* Confirmed diagnosis of active progressive multiple myeloma
* History of > 2 prior cytotoxic treatment regimens. Bone marrow transplantation will be considered as one regimen.
* Current measurable disease based on serum and/or urine M protein and/or measurable plasmacytoma.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
* Absolute neutrophil count (ANC) > 1,500 mm3
* Platelets > 100,000 mm3
* Serum creatinine < 1.5 upper limit of normal (ULN)
* Serum bilirubin < 1.5 ULN
* AST/AGOT and ALT/SGPT < 3.0 ULN
* Life expectancy > 12 weeks

Exclusion Criteria:

* Chemotherapy < 3 weeks prior to registration.
* Biologic or immunotherapy < 2 weeks prior to registration
* Full field radiotherapy < 4 weeks or limited field radiotherapy < 2 weeks prior to registration.
* History or presence of central nervous system (CNS) disease
* History of leukemia
* History of another primary malignancy with the exception of inactive basal or squamous cell carcinoma of the skin
* Major surgery < 4 weeks prior to registration
* Prior therapy with anti-vascular endothelial growth factor (VEGF) agents excluding thalidomide, Revimid, velcade and arsenic trioxide
* Interstitial pneumonia or extensive and symptomatic interstitial fibrosis of the lung
* Pleural effusion or ascites that cause respiratory compromise
* Female patients that are pregnant or breast feeding
* Uncontrolled high blood pressure, history of labile hypertension or history of poor compliance with an antihypertensive regimen
* Unstable angina pectoris
* Symptomatic congestive heart failure
* Myocardial infarction < 6 months prior to registration
* Serious uncontrolled cardiac arrhythmia
* Uncontrolled diabetes
* Active or uncontrolled infection
* Acute or chronic liver disease
* Impairment of gastrointestinal (GI) function or GI disease
* Confirmed HIV infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10
Dates: Start 2003-12; Primary Completion 2006-10 (Actual); Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
To determine the effectiveness of PTK in treating patients with relapsed or refractory myeloma

SECONDARY OUTCOMES:
To evaluate the progression free survival of patients treated with PTK
to investigate the safety of PTK in patients with relapsed/refractory multiple myeloma

CONTACTS AND LOCATIONS:
Overall Officials: Nikhil Munshi, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana-Farber Cancer Institute, Boston, Massachusetts, United States